CLINICAL TRIAL: NCT03252483
Title: A Randomized Controlled Trial to Evaluate Feasibility of Bundled HCV/HIV Rapid Screening
Brief Title: Integrating HIV and Hepatitis C Screening in an Urban Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Jason Leider, Director of Adult HIV Services, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2012-491
Record Dates: First submitted 2017-07-28; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C; Hiv; HIV/AIDS; HCV Coinfection; HIV/AIDS and Infections
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Infections | interventions — HIV Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV Only (Active Comparator): Those randomized to the control group were offered only an HIV test.
  Interventions: Other: HIV Screening
- Bundled HCV/HIV (Experimental): Those randomized to the intervention group were offered both HCV and HIV test.s
  Interventions: Other: Bundled HCV/HIV Screening

INTERVENTIONS:
Other: Bundled HCV/HIV Screening — Participants were randomized to a bundled HIV/HCV test group (intervention) to evaluate whether integrating HIV and HCV rapid screening would adversely impact HIV test acceptance.
  Arms: Bundled HCV/HIV
Other: HIV Screening — Participants were randomized to an HIV-only screening group as a control comparator.
  Arms: HIV Only

SUMMARY:
This randomized controlled trial was implemented to evaluate the effect of integrating rapid Hepatitis C (HCV) testing into a pre-existing screening program for Human Immunodeficiency Virus (HIV) on HIV test acceptance and diagnosis of both HCV and HIV. A sample of 478 adults in a New York City Emergency Department participated in the study. Participants were randomized to receive either an offer of bundled HIV/HCV testing or HIV testing alone. Public Health Advocates approached eligible patients in the Emergency Department, performed HIV and HCV raid testing, and delivered test results to participants with post-test counseling. The primary outcome, HIV test acceptance, was compared between the two groups to evaluate whether the addition of an HCV test adversely impacted participants' consent to test for HIV. Questionnaires were also distributed to participants to assess HCV knowledge.

DETAILED DESCRIPTION:
The high prevalence of HIV and HCV co-infection, similarity in testing strategies, and interrelated risk factors suggest a practical overlap in integrating screening services. This integration could effectively utilize existing resources and infrastructure to address both epidemics and facilitate the linkage of HCV-infected individuals to care.

The objective of this study was to integrate rapid HCV testing into a well-established HIV testing and counseling program to evaluate the effect of rapid bundled screening on HIV test acceptance rate. Secondary outcomes include HCV test acceptance, identification of newly diagnosed HCV- and HIV-positive patients, HCV knowledge, risk assessment, and refusal reasons.

The two-armed, randomized controlled trial was conducted at Jacobi Medical Center, a Level 1 trauma and tertiary care center located in the Bronx, New York. Upon recruitment, all participants completed questionnaires that included demographic information, HCV risk assessment, and HCV knowledge questions. Participants were randomized either to the control arm or the intervention arm. The control arm was offered HIV testing only and the intervention arm was offered HIV testing concurrently with HCV testing (bundled HIV/HCV screening).

Sample size was determined using the following parameters: 1) 80% power; 2) significance level of 0.05; 3) two-sided significant test; and 4) 10% difference between groups on the acceptance of HIV testing. Using these parameters, a sample of 227 in each group was needed to test the primary outcome: acceptance of an integrated screening program for HIV and HCV infection. Groups of at least 333 were used to allow for drop-outs and protocol violations.

Patients were recruited from the adult Emergency Department (ED) at Jacobi Medical Center. Recruitment took place during a six-month period from December 2012 to May 2013, and 478 patients were enrolled in the study.

Research Assistants were trained as Public Health Advocates to perform HIV and HCV testing and counseling. The Public Health Advocates approached eligible patients in the ED and followed a script to ask patients if they were interested in participating in a study through which they would be offered free screenings recommended for their general health. Patients who refused the offer of the HIV and/or HCV tests completed a test-refusal questionnaire. All enrolled participants completed a questionnaire including demographic information, HCV risk assessment, and HCV knowledge.

After providing verbal consent, participants were randomized to either an HIV test only group (control) or a bundled HIV/HCV test group (intervention). Randomization was performed by an independent statistician who used a computer generated allocation schedule. Randomization assignments were placed in sealed opaque envelopes that were opened sequentially after verbal consent was obtained for the study.

Those randomized to the control group were offered only an HIV test, and those randomized to the intervention group were offered both HCV and HIV tests. The OraQuick® HCV Rapid Antibody Test was employed as a rapid blood fingerstick test for HCV antibodies. The OraQuick Rapid Antibody Test Advance® HIV-1/2 Antibody test was used to test for HIV-1 and HIV-2 antibodies in oral fluid. Both point-of-care tests provide results in 20 minutes.

A Public Health Advocate delivered the test(s) results to the patient and conducted post-test counseling. In the case of a preliminary positive result on either test, the Public Health Advocate informed the patient and the patient's provider and scheduled a follow up appointment for the patient.

Data was recorded in an electronic database using Microsoft Excel (Microsoft Corp., Redmond, WA). Data obtained from subjects were entered using unique subject numbers, without specific identifiers. Acceptance rates for HIV testing in experimental and intervention arms was compared using chi square with fisher's exact derived confidence intervals. Stata statistical software was used to tabulate participant demographics and testing frequencies for HIV, HCV, or both.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Speak English or Spanish

Exclusion Criteria:

* Inability to consent
* Medically unstable as determined by healthcare provider
* Does not speak English or Spanish
* Known HIV and/or HCV positive
* Already tested for HIV and/or HCV within past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
HIV Test Acceptance | Through study completion, 6 months
  Participant agreement to test for HIV with a rapid Oraquick oral swab

SECONDARY OUTCOMES:
HCV Test Acceptance | Through study completion, 6 months
  Participant agreement to test for HCV with a rapid Orasure fingerstick
HIV and HCV Incidence | Through study completion, 6 months
  Diagnoses of either infection
HCV Knowledge and Risk | Through study completion, 6 months
  As assessed from a knowledge and risk assessment questionnaire distributed to each participant
Test Refusals | Through study completion, 6 months
  Reasons for refusal of either HIV or HCV tests

CONTACTS AND LOCATIONS:
Overall Officials: Jason Leider, MD, PhD, FACP, Study Chair — Jacobi Medical Center; Albert Einstein College of Medicine; New York City Health and Hospitals Corporation
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data includes HIV/HCV screening information and HCV knowledge and risk assessment. Study has been completed.